CLINICAL TRIAL: NCT04235686
Title: An 8 Week Randomized Double Blind Placebo Controlled Multi-site Study Assessing Efficacy and Safety of MYDAYIS® (D-amphetamine / L-amphetamine) for Bipolar Depression
Brief Title: 8 Week Multi-site Study of MYDAYIS® for Bipolar Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Lindner Center of HOPE (Other)
Responsible Party: Principal Investigator, Mark Frye, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-001722
Record Dates: First submitted 2019-12-04; First posted 2020-01-22 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Dextroamphetamine; Amphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study subjects will be randomized to receive MYDAYIS® or placebo on a 1:1 ratio according to computer-generated coding. Each site will have its own randomization list. Allocation concealment will be achieved by having the research pharmacy perform the randomization, package the study medication, and maintain the integrity of the blinded information throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mydayis - Active (Active Comparator): MYDAYIS®, Oral administration, dose regimen for Double blind phase and open label phase.
  12.5 mg x 7 days. 25 mg x 7 days 37.5 mg x 14 days 50 mg daily x 28 days
  Interventions: Drug: Mydayis Extended-Release Capsule
- Placebo (Placebo Comparator): Matching placebo, Oral administration, dose regimen for Double blind phase and open label phase.
  12.5 mg x 7 days. 25 mg x 7 days 37.5 mg x 14 days 50 mg daily x 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mydayis Extended-Release Capsule — Randomized, parallel - group, double-blind, placebo-controlled, flexible-dose adjunctive trial of MYDAYIS®
  Other Names: d-amphetamine / l-amphetamine
  Arms: Mydayis - Active
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This protocol is a Phase 2 multi-site study which aims to evaluate the safety and effectiveness of MYDAYIS® as adjunctive therapy for adults with bipolar depression. Results from this study WILL NOT be used to contribute to an approval of MYDAYIS ® for this indication.

ELIGIBILITY:
Inclusion Criteria

1. Male or female between 18 and 55 years of age
2. Bipolar I or II disorder as confirmed by structured diagnostic interview by Axis I of the SCID by DSM-IV-TR.
3. Currently experiencing a major depressive episode unresponsive to stable (i.e. at least 4 weeks) anti-manic mood stabilizers (lithium, valproate) and/or antipsychotic therapy, with or without concomitant antidepressant therapy.
4. Symptom severity score ≥11 on the self-report version of the Quick Inventory for Depressive Symptomatology (QIDS-SR16) or score ≥11 on the Quick Inventory for Depressive Symptomatology - Clinician (QIDS-C16) and ≥ 3 on the Clinical Global Impression for Bipolar Illness (CGI-BP) Depression Severity Scale.
5. Patients with a comorbid attention deficit disorder and binge eating disorder will be included.
6. Patients will be allowed to continue with their behavioral treatments (ie. CBT) targeted at their primary diagnosis.

Exclusion Criteria

1. Ability to provide informed consent and understand fully English and score ≥ 90% on comprehension test questionnaire that reviews study goals.
2. Clinically significant signs of suicidality from any of the following assessments:

   1. Response ≥ 4 on MADRS question # 10
   2. Response ≥2 on QIDS-C or QIDS-SR question # 12
   3. Yes response on Columbia Suicide Severity Scale (CSSR) Question # 3 (ideation without plan or intent) ,Question #4 (ideation with intent, but no plan), or Question # 5 (ideation, intent, and plan)
   4. Suicide attempt within the past year, as defined by the Columbia-Suicide Severity Scale
3. Known lifetime history of DSM-IV-TR diagnosis of cocaine or methamphetamine abuse or dependence. Nicotine dependence will be an exception.
4. Positive toxicology screen for drugs of abuse (ie. cocaine, methamphetamine, cannabis, opiates)
5. Known history of prescription abuse of stimulants.
6. Lifetime history of stimulant-induced mania
7. Active abuse or dependence of alcohol, opiates or cannabis that is either current or less than 3 months full remission.
8. Baseline Young Mania Rating Scale (YMRS) score ≥ 8
9. Patients with active psychosis identified by SCID or a diagnosis of schizophrenia, schizoaffective disorder, delusional or schizophreniform disorder.
10. Known hypersensitivity, such as angioedema or anaphylaxis, to amphetamines or other ingredients of MYDAYIS.
11. Clinically unstable medical disease
12. Known history of a structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormality, coronary artery disease, stroke or other serious cardiovascular problems.
13. ECG with significant arrhythmias, conduction abnormalities, or voltage criteria met for left ventricular hypertrophy (unless cleared by cardiology consultation).
14. Uncontrolled hypertension (>160/100) or tachycardia (heart rate >110)
15. History of grand mal seizure; history of febrile seizure as infant permitted
16. Established vasculopathy or history of Raynaud's phenomena
17. Narrow angle glaucoma
18. Patients with end stage renal disease (ESRD).
19. Concomitant treatment with monoamine oxidase inhibitors (MAOIs), and also within 14 days following discontinuation of treatment with a monoamine oxidase inhibitor.
20. Tourette's syndrome
21. Women who are pregnant, lactating or of child-bearing potential and not using at least one adequate contraceptive measure (i.e. hormonal contraception-birth control pills-, intrauterine devices (IUD), tubal ligation or condoms during sexual intercourse)
22. Men who do not use adequate measures (male condoms).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) score | Baseline to week 8 visit 10
  Reduction in Montgomery-Asberg Depression Rating Scale (MADRS) score (Range: 0-60) between Baseline and Week 8 visit 10

SECONDARY OUTCOMES:
Change in Quick Inventory for Depressive Symptomatology (QIDS-C and QIDS-SR) score | Baseline to Week 8 visit 10
  Reduction in Clinician and self-report symptoms of depression as measured by the Quick Inventory for Depressive Symptomatology (QIDS-C and QIDS-SR) (Range: 0-27)
Remission | Baseline to Week 8 visit 10
  Treatment remission (Montgomery-Asberg Depression Rating Scale (MADRS) score < 10) (Range 0-60)
Change in General Anxiety Disorder 7-item scale score | Baseline to Week 8 visit 10
  Self-report anxiety as measured by the General Anxiety Disorder 7-item scale (GAD-7) (Range: 0-21)
Response | Baseline to Week 8 visit 10
  Treatment response (50% reduction in Montgomery-Asberg Depression Rating Scale (MADRS) score (Range: 0-60)
Change in Clinical Global Impression for Bipolar Disorder (CGI-BP) score | Baseline to Week 8 visit 10
  Percentage of much or very much improved as measured by the Clinical Global Impression for Bipolar Disorder (CGI-BP) (Range: 1-8)
Change in Young Mania Rating Scale (YMRS) score | Baseline to Week 8 visit 10
  Reduction in sub-syndromal manic symptoms as measured by the Young Mania Rating Scale (YMRS) (Range: 0-56)
Change in Epworth Sleepiness Scale (ESS) score | Baseline to Week 8 visit 10
  Self-report likelihood of falling asleep during normal daily situations as measured by the Epworth Sleepiness Scale (ESS) (Range: 0-24)
Change in Fatigue Severity Scale (FSS) score | Baseline to Week 8 visit 10
  Self-report measure of fatigue as measured by the Fatigue Severity Scale (FSS) (Range: 0-63)
Change in Binge Eating Scale (BES) score | Baseline to Week 8 visit 10
  Self-report binge eating behavior as measured by the Binge Eating Scale (BES) (Range: 0-48)
Change in Morningness-Eveningness Questionnaire (MEQ) score | Baseline to Week 8 visit 10
  Self-Report measure on the Morningness-Eveningness Questionnaire (MEQ) (Range: 16-86)
Change in Rapid Eating and Activity Assessment for Patients (REAP) score | Baseline to Week 8 visit 10
  Self-Report measure on Rapid Eating and Activity Assessment for Patients (REAP) (Range: 0-27)
Change in Digit Symbol Substitution Test (DSST) score | Baseline to Week 8 visit 10
  Improvement in cognition as measured by the Digit Symbol Substitution Test (DSST) (Range: 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Frye, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Lindner Center of Hope, Mason, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials